CLINICAL TRIAL: NCT02239159
Title: Acupuncture-assisted-anesthesia to Improve Complications After Digestive Surgery in Elderly Patients:Multi-center Double-blinded Randomized Controlled Trial
Brief Title: Acupuncture-assisted-anesthesia to Improve Postoperative Outcome After Digestive Surgery in Elderly Patients
Acronym: AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr., Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-2014-02-21-1
Record Dates: First submitted 2014-04-06; First posted 2014-09-12 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Complications; Surgery
Keywords: transcutaneous electric acupoint stimulation; elderly patients
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Electrodes will be attached, but stimulation will not be given
- Non-acupoint TES (Sham Comparator): TES is for transcutaneous electric stimulation.Stimulation will be given through electrodes attached to non-acupoints
  Interventions: Other: TES(transcutaneous electric stimulation)
- Acupoint TES (Experimental): Transcutaneous stimulation will be given through acupoints
  Interventions: Other: TES(transcutaneous electric stimulation)

INTERVENTIONS:
Other: TES(transcutaneous electric stimulation) — Stimulation will be given through electrodes attached to the skin
  Arms: Acupoint TES; Non-acupoint TES

SUMMARY:
The investigators assume that transcutaneous electric acupoint stimulation (TEAS) pretreatment may activate the endogenous protective mechanism, as a result protect the patients against subsequent surgical stress pregnancy. And TEAS may induce the production of endogenous analgesic transmitters, so develop an anesthetic-sparing effect. The investigators believe this intervention will reduce the subsequent incidence, duration and severity of organ dysfunction, possibly reducing the morbidity, even mortality. So in this study, the investigators hypothesize that TEAS before anesthesia and during surgery would decrease the morbidity and mortality of postoperative complications in 30 days after digestive surgery in elderly patients .

DETAILED DESCRIPTION:
Patients older than 65 years old are at higher risk of postoperative morbidity and mortality. With the increasing number of old patients scheduled for digestive surgery, exploring methods to decrease postoperative morbidity is very important. Noninvasive methods may be easier to clinically use. Transcutaneous electric acupoint stimulation (TEAS)has been proved to decrease need for general anesthetics during anesthesia, and to alleviate systemic inflammatory response. Considering the morbidity and mortality after surgery is closely related to use of anesthetics and inflammatory response,TEAS may be a good selection for improving postoperative outcomes.Among the postoperative complications, pulmonary complication and systemic inflammatory response syndrome is with higher incidence, so we will focus on these two complications in our study.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Age ≥65 years of age
* Elective digestive surgery under general anesthesia

Exclusion Criteria:

* ASA(American Society of Anesthesiologists) status> Ⅲ
* Patients undergoing surgery within 12 h of admission to hospital
* Patients undergoing surgery of the chest
* Patients suffered from neurologic disorder or impaired mental state
* Patients with contraindications to the use of electro-acupuncture, such as skin damage or infection at the acupoints
* Patients with experience of transcutaneous electrical stimulation treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 748 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Pulmonary Adverse Events as a Measure of Morbidity Tolerability | participants will be followed from the end of the surgery to 30 days after surgery

SECONDARY OUTCOMES:
Number of participants died of all causes | Participants will be followed from the end of the surgery to 30 days after surgery
Length of ICU stay | participants will be followed for the duration of hospital stay after surgery, an expected average of 7 days
Number of participants with ICU admission | participants will be followed for the duration of hospital stay after surgery, an expected average of 7 days
Number of participants with Systemic Inflammatory Response Syndrome(SIRS) | Participants will be followed from the end of the surgery to 30 days after surgery
Length of hospital stay | participants will be followed for the duration of hospital stay after surgery, an expected average of 7days

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, PhD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital,Fourth Military Medical University, Xi'an, Shaanxi, China